CLINICAL TRIAL: NCT03425084
Title: Genetic Variation in Organic Cation Transport 1 (OCT1) and Its Significance for Morphine Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Council for Independent Research (Other); The Faculty of Health Sciences SDU (Unknown); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ida Kuhlmann, MD, phd student, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AKF-391
Record Dates: First submitted 2018-01-15; First posted 2018-02-07 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2018-01

CONDITIONS: Organic Cation Transporter 1; Morphine
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morphine (Experimental): Intravenous morphine (0,15 mg/kg) will be given as a single dosis at the end of the surgery followed by morphine administrated by patient-controlled analgesia (PCA) as single boluses (0,04mg/kg)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — The study was designed as an open, non-controlled drug trial, with scientists and participants blinded to the patients OCT1 status. Morphine will be given as a single dosis (0,15 mg/kg) at the end of the Surgery and later as boluses of 0,04mg/kg administrated by patient-controlled analgesia, (PCA). Blood samples with drug concentrations will be used to determine a difference in morphine AUC due to the patients OCT1 status. Questionnaire answers will be used to determine the effect of morphine due to the patients OCT1 status

SUMMARY:
The main objective of the trial is to investigate the effect of known genetic variants in organic cation transporter 1 (OCT1) on the effect of morphine after major surgery

DETAILED DESCRIPTION:
The purpose of the experiment is to investigate the effect of known genetic variants in organic cation transporter 1 (OCT1) on the effect of morphine after major surgery. This is primarily done by investigating systemic exposure of morphine in a cohort of patients undergoing scheduled laparoscopic colon or laparoscopic rectum surgery, and as pain treatment with intravenous (iv) morphine at the end of and after surgery (primary endpoints). As a secondary endpoint, we will investigate the effect (pharmacodynamics) of morphine in the same patients by registering pain during rest and activity, side effects and the degree of sedation at appropriate time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Planned Colectomy / Hemicolectomy, sigmoid resection, rectal resection or abdominal perianal amputation of the rectum with stoma, good general health (ASA 1 -2), Informed consent given, Age 18-90 years and BMI 18,5 - 35kg/m².

Exclusion Criteria:

* Abdominoperineal resection (APR) - ad modum Holm (abdominal perianal amputation of rectum with stoma)
* Daily use of opioids
* Indicator for the use of an epidural catheter
* Alcohol abuse
* Hypersensitivity for morphine
* A known serious disease (Terminal cancer, severe dementia, significant heart, liver, lung or renal failure or severe psychiatric disease)
* Women of childbearing age who do not use safe contraception
* Women who are breastfeeding
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Morphine Area under the curve (AUC) | Blood samples will be drawn at zero, five, 10, 15, 30, 45, 60 and 90 minutes after the first morphine bolus
  Difference in morphine AUC due to patient OCT1 status

SECONDARY OUTCOMES:
Morphine effect | Questionnaire answers will be collected with an appropriate time interval for 24 hours after the first morphine bolus
  Pain during rest and activity will be evaluated through a Numeric Rating Scale on the same patients where 0 is no pain and 10 is the the worst possible pain.
Morphine effect | Questionnaire answers will be collected with an appropriate time interval for 24 hours after the first morphine bolus
  side effects will be evaluated through a 5-point verbal questionnaire on the same patients where 0 is no side effects and 4 is unacceptable side effects.
Morphine effect | Questionnaire answers will be collected with an appropriate time interval for 24 hours after the first morphine bolus
  The degree of sedation will be evaluated through the Richmond Agitation and Sedation Scale (RASS) on the same patients
Morphine effect | After the trial has ended (24 hours after the first morphine bolus) data containing morphine use will be collected.
  The total dose of morphine used during the investigation.
Morphine effect | After the trial has ended (24 hours after the first morphine bolus) data containing morphine use will be collected.
  The number of administrations of morphine will be recorded

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Sydvestjysk Sygehus, Esbjerg
  - Odense Universitetshospital, Odense